CLINICAL TRIAL: NCT07186296
Title: EXoPERT EMERALD: Early Multi-cancer Study of EV's Ramen-AL Linked Diagnosis Clinical Study Protocol
Brief Title: EXoPERT EMERALD Clinical Study
Status: Recruiting | Type: Observational
Sponsor: EXoPERT (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Other Study IDs: EXPT-MC-F-2024
Record Dates: First submitted 2025-08-29; First posted 2025-09-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Colon Cancer; Pancreatic Cancer; Ovarian Cancer; Lung Cancer
Keywords: Early-stage; In vitro Diagnostic Test; Artificial intelligence; extracellular vesicles; multi cancer diagnosis; cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Prospective with frozen plasma aliquots being retained. Frozen exosomes are also being stored after testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (6):
- Control
  Interventions: Diagnostic Test: EXoPred
- Lung Cancer
  Interventions: Diagnostic Test: EXoPred
- Breast Cancer
  Interventions: Diagnostic Test: EXoPred
- Colorectal Cancer
  Interventions: Diagnostic Test: EXoPred
- Pancreatic Cancer
  Interventions: Diagnostic Test: EXoPred
- Ovarian Cancer
  Interventions: Diagnostic Test: EXoPred

INTERVENTIONS:
Diagnostic Test: EXoPred — Performing invitro Diagnostics with devices developed by EXoPERT.

SUMMARY:
Invitro diagnostic test for multiple cancer diagnosis for patients with early-stage cancers by analyzing surface-enhanced Ramen spectroscopy (SERS) profiles of extracellular vesicles (EV) using artificial intelligence.

DETAILED DESCRIPTION:
An in vitro diagnostic medical device and system that provides information on the presence of lung, ovarian, breast, pancreas and colorectal cancers based on a deep learning analysis for Raman spectroscopic profiles of EV's extracted from human plasma. Tissue of origin (TOO) can be presented as one or more.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 45 years or older with a biopsy-proven or clinically suspected primary lung, breast, colorectal, pancreatic, or ovarian cancer, based on objective findings such as radiological, serological, endoscopic, or cytological findings, whose blood was collected prior to any systemic or definitive therapy for the cancer.
* Subjects who are willing and able to provide written informed consent.
* Subjects who are willing and able to comply with the study requirements.

Exclusion Criteria:

* Any history of cancer diagnosed and treated within 5 years prior to the date of consent.
* Subjects with a history of previous cancer treatment via surgical resection, hormonal cancer treatment, chemotherapy, radiotherapy within the past 6 months for recent cancer diagnosis.
* Subjects who have any history of an allogeneic bone marrow, stem cell transplant, or solid organ transplant.
* Subjects who are pregnant or breastfeeding women.
* Subjects who have consented and have undergone treatment in any other cancer related clinical trials withinthe past 6 months.
* Subjects who are currently in active treatment for drug abuse.
* Subjects who have received any treatment related to lung, breast, colorectal, pancreatic, or ovarian nodules, such as hormones prior to entering the study.
* Unsuitable sample for testing due to contamination, hemolysis, etc.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be collected from hospitals/clinical care settings with access to the intended population.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Test Sufficient Samples | From date of enrollment up to 36 months
  Test sufficient samples from 5 cancers to lock an validate algorithm to support future clinical study.
Evaluate Performance | From date of enrollment up to 36 months
  Test performance: diagnosis of multiple cancer, assessed by sensitivity. Test performance: diagnosis of multiple cancer, assessed by specificity. Test performance: diagnosis of multiple cancer, assessed by tissue of origin (TOO) accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dudley, MD, Principal Investigator — Johns Hopkins University; Saeed Jortani, Ph.D., Principal Investigator — Kentucky Clinical Trial Laboratory
Locations (9):
- United States (9):
  - Tibor Rubin VA Medical Center, Long Beach, California
  - City of Hope Duarte Cancer Center, Los Angeles, California
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Lexington VA Healthcare System, Lexington, Kentucky
  - KCTL, Louisville, Kentucky
  - John Hopkins University, Baltimore, Maryland
  - Albany Stratton VA Medical Center, Albany, New York
  - Bronx Veterans Medical Research Foundation, The Bronx, New York
  - VA Hudson Valley Healthcare System, Wappingers Falls, New York

IPD SHARING:
Plan to Share IPD: Undecided